CLINICAL TRIAL: NCT01314560
Title: Study of the Pathophysiological Mechanisms Involved in Bleeding Events Observed in Patients With Lowe Syndrome
Brief Title: Study of the Pathophysiological Mechanisms Involved in Bleeding Events
Acronym: LOWE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P071008
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Oculocerebrorenal Syndrome
Keywords: Lowe syndrome; OCRL; Haemostasis; Bleeding Disorders; Platelet Function Tests
MeSH Terms: conditions — Oculocerebrorenal Syndrome; Hemostatic Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): experimental
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample

SUMMARY:
Lowe syndrome is associated with mutations in the OCRL1 gene, which encodes OCRL1, a phosphatidylinositol-4, 5-bisphosphate (PtdIns(4, 5)P (2))5-phosphatase. PtdIns(4, 5)P2, a substrate of OCRL1, is an important signaling molecule within the cell. An abnormal rate of hemorrhagic events was found in a retrospective clinical survey, suggesting platelet dysfunction.

The main objective of the study is to confirm the presence of platelet dysfunction in Lowe syndrome and to characterize this abnormality.

DETAILED DESCRIPTION:
Introduction: Lowe syndrome (LS), also known as oculocerebrorenal syndrome of Lowe (OCRL), is a rare X-linked condition characterized by congenital cataracts, defective renal tubule cell function, muscular hypotonia and variable degrees of mental retardation. Patients with LS require frequent surgery, some of which are associated with a severe haemorrhagic risk, such as scoliosis reduction, hip surgery, or eye surgery. In a recent retrospective clinical survey of French LS patients, we observed an abnormal rate of haemorrhagic events, some of which had dramatic outcomes. LS is caused BYMUTATIONS in the OCRL gene, which encodes OCRL, an inositol polyphosphate 5-phosphatase. The preferred OCRLsubstrate is the membrane phospholipid phosphatidylinositol-4,5-bisphosphate (PtdIns(4,5)P2). OCRL also contains a Rho GTPase-activating protein(GAP)-like domain that participates in the regulation of Rho proteins (Rho, Rac, Cdc42), as GTPase-activating proteins or by mediating in protein-protein interactions. PtdIns(4,5)P2 and Rho-dependent signalling play a central role in many important cellular processes, including vesicular trafficking and cytoskeletal organization both of which are very important for platelet function. Thus, modulation of PtdIns(4,5)P2 levels and/or Rho-dependent signalling would be expected to impact platelet function.

Based on the clinical observation, we tested whether hemorrhagic symptom of 6 Lowe patients could be related to homeostasis abnormalities and we found that all the six patients had a prolonged closure time tested by PFA100 analyzer (Platelet Function Analyzer). These results were measured in absence of interfering factor such anemia, thrombopenia, or von Willebrand factor deficiency, thus suggesting platelet dysfunction.

Study justification:

The comprehension of the physiopathology implicated in the abnormal hemorrhagic risk is of major interest in term of prevention and clinical management in Lowe patients who requires frequent surgical care.

Objectives:

The main objective of the study is to confirm the presence of platelet dysfunction in Lowe syndrome and to characterize this abnormality. The secondary aims are to settle a functional test allowing the detection of patients with increasing hemorrhagic risk. Moreover, we could determinate whether platelet is an interesting cellular model, easily available, for further OCRL1 studies in Lowe patients.

Methods:

We will investigate platelet activation response in 15 Lowe cases and 15 normal cases. The evaluation criteria will include the PFA100, THROMBOELASTOMETRY (ROTEM), aggregation, secretion, adhesion in a flux system and clot retraction. We will also compare molecular (phospho-proteins, phospholipid...) and structural modifications of the non activated platelet and of activating platelet.

Conclusion:

The characterization of a platelet activation abnormality in Lowe patients could lead to major benefit for the patients with systematic homeostasis screening and special precautions rules before surgery, often required in this multisystemic condition. Moreover, this study could contribute to go further into PI(4,5)P2 signaling pathways and may provide clues to the interrelationship between these processes in normal metabolism and diseases states.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a clinical syndrome of Lowe (congenital cataracts, renal tubular dysfunction and neuromuscular damage) with a molecular defect in the gene known OCRL1.
* For the centre of Necker, patients should have a weight> 10 kg. For the centre of Toulouse site, patients should have a weight> 40 kg.
* No alteration of glomerular function (creatinine clearance> 30 ml/min/1.73m ²)
* No significant anemia (hematocrit> 25%, hemoglobin> 8 g / L)
* Every patient should have included a signed informed consent. For minor patients, the consent of parents or legal guardian must be obtained.
* Patients may be included only if they receive social security coverage or CMU

Exclusion Criteria:

* Weight less than 10 kg for the centre of Necker
* Weight less than 40 kg for the centre of Toulouse
* Major renal insufficiency (creatinine clearance <30 ml/min/1.73m ²)
* Profound anemia (hematocrit <25%, Hb <8g/dl)
* Patients taking drugs interfering with hemostasis in the eight days before the survey
* Patients with major behavior disorder making it difficult to achieve the blood sample, despite the nitrous oxide
* Patients with a other pathology of hemostasis (hemophilia, thrombotic disease)
* Participation in another clinical study requiring a blood sample within 4 weeks
* Contraindication to EMLA patch: confers Summary of Product Characteristics.
* Contraindication to KALINOX: confers Summary of Product Characteristics.

Ages: 6 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The platelet function will be evaluated by comparing the intensity of platelet responses obtained in patient and controls | 18 months
  The platelet function will be evaluated by comparing the intensity of platelet responses obtained in patient and controls. Various platelet responses will be studied:
  * The measurement of platelet closure time by PFA100
  * Aggregation, retraction, secretion and adhesion

SECONDARY OUTCOMES:
Characterization of abnormalities in platelet-signalling pathways | 18 months
  Characterization of abnormalities in platelet-signalling pathways

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Baujat, MD, PhD, Principal Investigator — Hôpital Necker Enfants Malades, Paris
Locations (1):
- Necker Enfants Malades Hospital, Genetic, Paris, France

REFERENCES:
- [Result] Egot M, Lasne D, Poirault-Chassac S, Mirault T, Pidard D, Dreano E, Elie C, Gandrille S, Marchelli A, Baruch D, Rendu J, Faure J, Flaujac C, Gratacap MP, Sie P, Gaussem P, Salomon R, Baujat G, Bachelot-Loza C. Role of oculocerebrorenal syndrome of Lowe (OCRL) protein in megakaryocyte maturation, platelet production and functions: a study in patients with Lowe syndrome. Br J Haematol. 2021 Mar;192(5):909-921. doi: 10.1111/bjh.17346. Epub 2021 Feb 2. PMID 33528045